CLINICAL TRIAL: NCT03004638
Title: A Phase 2a Randomized, Blinded, Placebo-controlled Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Multiple Ascending Doses of MEDI6012 in Subjects With Stable Atherosclerotic Cardiovascular Disease
Brief Title: Multiple Ascending Doses of MEDI6012 in Subjects With Stable Atherosclerotic Cardiovascular Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5780C00005
Record Dates: First submitted 2016-12-12; First posted 2016-12-29 (Estimated); Results first posted 2018-11-30 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Atherosclerosis; Cardiovascular Disease
Keywords: Atherosclerosis; Cardiovascular Disease; CAD; Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- MEDI6012 40 mg (Experimental): Participants received 3 doses of 40 milligram (mg) MEDI6012 IV on Days 1, 8, and 15.
  Interventions: Drug: MEDI6012 40 mg
- Placebo (Placebo Comparator): Participants received 3 doses of placebo matching with MEDI6012 intravenously (IV) on Days 1, 8, and 15.
  Interventions: Drug: Placebo
- MEDI6012 120 mg (Experimental): Participants received 3 doses of 120 mg MEDI6012 IV on Days 1, 8, and 15.
  Interventions: Drug: MEDI6012 120 mg
- MEDI6012 300 mg (Experimental): Participants received 3 doses of 300 mg MEDI6012 IV on Days 1, 8, and 15.
  Interventions: Drug: MEDI6012 300 mg
- MEDI6012 IV Push (Experimental): Participants received 3 doses of MEDI6012 by IV push as 300 mg loading dose on Day 1, and maintenance doses of 150 mg and 100 mg on Day 3 and Day 10, respectively.
  Interventions: Drug: MEDI6012 IV Push
- Placebo IV Push (Placebo Comparator): Participants received 3 doses of placebo matching with MEDI6012 by IV push. A loading dose on Day 1 and maintenance doses on Days 3 and 10.
  Interventions: Drug: Placebo IV Push

INTERVENTIONS:
Drug: MEDI6012 40 mg — Participants received 3 doses of 40 milligram (mg) MEDI6012 IV on Days 1, 8, and 15.
  Arms: MEDI6012 40 mg
Drug: Placebo — Participants received 3 doses of placebo matching with MEDI6012 intravenously (IV) on Days 1, 8, and 15.
  Arms: Placebo
Drug: MEDI6012 120 mg — Participants received 3 doses of 120 mg MEDI6012 IV on Days 1, 8, and 15.
  Arms: MEDI6012 120 mg
Drug: MEDI6012 300 mg — Participants received 3 doses of 300 mg MEDI6012 IV on Days 1, 8, and 15.
  Arms: MEDI6012 300 mg
Drug: Placebo IV Push — Participants received 3 doses of placebo matching with MEDI6012 by IV push. A loading dose on Day 1 and maintenance doses on Days 3 and 10.
  Arms: Placebo IV Push
Drug: MEDI6012 IV Push — Participants received 3 doses of MEDI6012 by IV push as 300 mg loading dose on Day 1, and maintenance doses of 150 mg and 100 mg on Day 3 and Day 10, respectively.
  Arms: MEDI6012 IV Push

SUMMARY:
To evaluate the safety pharmacokinetics, and pharmacodynamics of repeat weekly dosing of MEDI6012 in subjects with stable atherosclerosis.

DETAILED DESCRIPTION:
A Phase 2a Randomized, Blinded, Placebo-controlled Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Doses of MEDI6012 in Subjects with Stable Atherosclerotic Cardiovascular Disease

ELIGIBILITY:
Inclusion Criteria:

* Non-childbearing potential
* Diagnosis of stable atherosclerotic CVD
* Currently receiving a stable dose of Statin

Exclusion Criteria:

* Unstable cardiovascular condition within 3 months of screening
* Elective arterial revascularization with in the past month
* Any planned arterial revascularization
* Body mass index <18 or >45
* Clinically significant ECG that may interfere with the interpretation of serial ECG and QT interval changes at screening
* Chronic kidney disease defined by estimated glomerular filtration rate of less than 30 mL/mim/1.73m2
* Triglycerides greater than 500 mg/dL, LDL-C greater than 160 mg/dL, or HDL-C greater than 60 for males, or 65 for females
* Clinically significant vital sign abnormalities
* Genetic disorder of cholesterol metabolism
* History of overt liver disease
* Poorly controlled endocrine disorder (Diabetes or Thyroid disorder)
* Current or recent use of systemic corticosteroids
* Recent or ongoing infection or febrile illness
* History of active malignancy within 5 years
* History of alcohol or recreational substance abuse in the past 6 months
* Concurrent enrollment in another clinical study of any investigational drug therapy or use of any biologicals within 6 months prior to screening or within 5 half-lives of an investigational agent or biologic, whichever is longer.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Research Site, Anniston, Alabama
  - Research Site, Jacksonville, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Cincinnati, Ohio

REFERENCES:
- See also: D5780C00005-CSP-amendment-1_REDACTED_16Jul2017_PDF-A — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4211&filename=D5780C00005-CSP-amendment-1_REDACTED_16Jul2017_PDF-A.pdf
- See also: 5780C00005 MEDI6012 Statistical Analysis Plan_21Jul2017_Version2_Redacted_PDF-A.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4211&filename=5780C00005%20MEDI6012%20Statistical%20Analysis%20Plan_21Jul2017_Version2_Redacted_PDF-A.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 4 sites in the USA between 23Jan2017 and 02Nov2017.
Pre-assignment Details: A total of 91 participants were screened, of which 32 participants were randomized in a 6:2 ratio to receive MEDI6012 or placebo in 4 cohorts (8 participants in each cohort). For Cohort 4, randomization happened in a 7:1 ratio to receive MEDI6012 or placebo due to an interactive voice/web response system programming issue.
Period: Overall Study
Arm/Group | Placebo | MEDI6012 40 mg | MEDI6012 120 mg | MEDI6012 300 mg | Placebo IV Push | MEDI6012 IV Push
Started | 6 | 6 | 6 | 6 | 1 | 7
Completed | 6 | 6 | 6 | 6 | 1 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received at least one dose of study drug.
Groups:
- Cohort 1: MEDI6012 40 mg: Participants received 3 doses of 40 milligram (mg) MEDI6012 IV on Days 1, 8, and 15.
- Cohort 2: MEDI6012 120 mg: Participants received 3 doses of 120 mg MEDI6012 IV on Days 1, 8, and 15.
- Cohort 3: MEDI6012 300 mg: Participants received 3 doses of 300 mg MEDI6012 IV on Days 1, 8, and 15.
- Cohort 4: MEDI6012 IV Push: Participants received 3 doses of MEDI6012 by IV push as 300 mg loading dose on Day 1, and maintenance doses of 150 mg and 100 mg on Day 3 and Day 10, respectively.
- Total: Total of all reporting groups
Arm/Group | Placebo | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Placebo IV Push | Cohort 4: MEDI6012 IV Push | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 1 | 7 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.8 (4.8) | 66.7 (3.3) | 68.8 (2.8) | 66.2 (2.6) | 65.0 (NA) — Standard deviation was not applicable as only one participant was evaluable for this reporting group. | 71.4 (4.2) | 68.2 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 3 | 0 | 1 | 9
  Male | 4 | 4 | 5 | 3 | 1 | 6 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 1 | 0 | 3
  White | 5 | 6 | 6 | 5 | 0 | 7 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 6 | 6 | 6 | 1 | 7 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience(immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are the events between first dose of study drug and up to 56 days after last dose of study drug (Day 66 for Cohort 4 and placebo IV push arm and Day 71 for Cohorts 1 to 3 and placebo arm) that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: From Day 1 to Day 56 after last dose of study drug (Day 66 for Cohort 4 and Placebo IV push arm and Day 71 for Cohorts 1 to 3 and placebo arm)
Population: As-treated population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Placebo IV Push | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 1 | 7
Participants
  TEAEs | 3 | 3 | 3 | 4 | 0 | 3
  TESAEs | 0 | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Evaluations Reported as TEAEs
Description: An abnormal laboratory finding which required an action or intervention by the investigator, or a finding judged by the investigator as medically significant was reported as an AE. Laboratory evaluations included haematology, serum chemistry, and urinalysis.
Time Frame: as for outcome 1
Population: As-treated population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Placebo IV Push | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 1 | 7
Participants | 0 | 1 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: Treatment-emergent adverse events observed in participants with clinically significant vital signs abnormalities are reported. Vital sign parameters included blood pressure, respiration rate, heart rate, pulse oximetry, and body temperature.
Time Frame: as for outcome 1
Population: As-treated population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Placebo IV Push | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 1 | 7
Participants
  Hypertension | 1 | 1 | 0 | 0 | 0 | 0
  Hypotension | 0 | 0 | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Abnormal Electrocardiogram Reported as TEAEs
Description: Treatment-emergent adverse events observed in participants with clinically significant ECG abnormalities are reported.
Time Frame: as for outcome 1
Population: As-treated population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Placebo IV Push | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 1 | 7
Participants | 0 | 0 | 1 | 0 | 0 | 0

5. Primary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hour (hr) (AUC [0-96 hr]) Post Dose 3 for High-density Lipoprotein-cholesterol (HDL-C)
Description: The AUC (0-96 hr) is the area under the concentration-time curve from time 0 to 96 hrs of high-density lipoprotein-cholesterol.
Time Frame: Pre-dose, end of infusion, 12, 24, and 96 hrs post Day 15 dose (third dose) for Cohorts 1 to 3 and Placebo arm; Pre-dose, end of infusion, 12, 24, and 96 hrs post Day 10 dose (third dose) for Cohort 4 and Placebo IV push arm.
Population: As-treated population included all participants who received at least one dose of study drug. The overall number of participants analyzed denotes the number of participants evaluated specific for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg*h/dL
Arm/Group | Placebo | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Placebo IV Push | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 1 | 7
mg*h/dL | -6.72 (467.59) | 1355.64 (576.94) | 2874.86 (1232.21) | 6465.05 (2074.77) | 266.68 (NA) — Standard deviation was not applicable as only one participant was evaluable for this reporting group. | 1803.12 (1684.32)

6. Primary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hour (hr) (AUC [0-96 hr]) Post Dose 3 for High-density Lipoprotein-cholesterol Ester (HDL-CE)
Description: The AUC (0-96 hr) is the area under the concentration-time curve from time 0 to 96 hrs of high-density lipoprotein-cholesterol ester.
Time Frame: as for outcome 5
Population: As-treated population included all participants who received at least one dose of study drug.The overall number of participants analyzed denotes the number of participants evaluated specific for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg*h/dL
Arm/Group | Placebo | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Placebo IV Push | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 1 | 7
mg*h/dL | -23.75 (422.76) | 1161.47 (506.67) | 2580.51 (1076.11) | 5710.09 (1622.36) | 273.03 (NA) — Standard deviation was not applicable as only one participant was evaluable for this reporting group. | 1597.12 (1531.40)

7. Primary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hour (hr) (AUC [0-96 hr]) Post Dose 3 for Cholesterol Ester
Description: The AUC (0-96 hr) is the area under the concentration-time curve from time 0 to 96 hrs of cholesterol ester.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg*h/dL
Arm/Group | Placebo | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Placebo IV Push | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 1 | 7
mg*h/dL | 373.04 (1060.76) | 2267.37 (1126.43) | 4047.38 (1314.67) | 9004.31 (2086.47) | 371.75 (NA) — Standard deviation was not applicable as only one participant was evaluable for this reporting group. | 2649.56 (3039.83)

8. Secondary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hour (hr) (AUC [0-96 hr]) Post Dose 3 for Apolipoprotein A1
Description: The AUC (0-96 hr) is the area under the concentration-time curve from time 0 to 96 hrs of Apolipoprotein A1.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg*h/dL
Arm/Group | Placebo | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Placebo IV Push | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 1 | 7
mg*h/dL | 821.33 (1465.70) | 2440.48 (1021.34) | 3740.59 (1508.93) | 5302.87 (1739.86) | -20.42 (NA) — Standard deviation was not applicable as only one participant was evaluable for this reporting group. | 2399.42 (2611.21)

9. Secondary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hour (hr) (AUC [0-96 hr]) Post Dose 3 for Low-density Lipoprotein Cholesterol (LDL-C).
Description: The AUC (0-96 hr) is the area under the concentration-time curve from time 0 to 96 hrs of LDL-C.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg*h/dL
Arm/Group | Placebo | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Placebo IV Push | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 1 | 7
mg*h/dL | -55.96 (886.81) | 1125.45 (872.40) | 1043.39 (700.00) | 3056.76 (1765.33) | -78.79 (NA) — Standard deviation was not applicable as only one participant was evaluable for this reporting group. | 1364.12 (2375.93)

10. Secondary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hour (hr) (AUC [0-96 hr]) Post Dose 3 for Apolipoprotein B
Description: The AUC (0-96 hr) is the area under the concentration-time curve from time 0 to 96 hrs of Apolipoprotein B.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg*h/dL
Arm/Group | Placebo | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Placebo IV Push | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 1 | 7
mg*h/dL | -82.95 (667.65) | -40.06 (477.21) | 145.42 (283.62) | -374.38 (588.54) | -239.17 (NA) — Standard deviation was not applicable as only one participant was evaluable for this reporting group. | 73.01 (864.30)

11. Secondary Outcome: Change From Baseline in Serum Concentration for MEDI6012 Mass
Description: The trough concentration level of MEDI6012 following each dose is reported (concentration at Days 8, 15, and 22 for Cohorts 1 to 3 and placebo; Concentration at Days 3, 10, and 17 for Cohort 4 and placebo IV push arm).
Time Frame: Seven days post-dose following Doses 1 to 3 in Cohorts 1 to 3 and placebo arm (Days 8, 15, 22); 2 days post-dose following Dose 1 (Day 3) and 7 days post-dose following Doses 2 and 3 (Days 10, 17) in Cohort 4 and placbo IV push.
Population: Pharmacokinetic (PK) population included all participants in the as-treated population who had at least one detectable lecithin-cholesterol acyltransferase (LCAT) serum concentration measurement. The overall number of participants analyzed denotes the number of participants evaluated specific for this outcome measure.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Placebo | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Placebo IV Push | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 1 | 7
μg/mL
  Day 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 7
  Day 3 |  |  |  |  | 0.0000 (NA) — Standard deviation was not applicable as only one participant was evaluable for this reporting group. | 16.2684 (4.5094)
  Day 8: number analyzed (Participants) | 6 | 6 | 6 | 5 | 0 | 0
  Day 8 | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 3.8646 (2.0753) |  |
  Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 7
  Day 10 |  |  |  |  | 0.0000 (NA) — Standard deviation was not applicable as only one participant was evaluable for this reporting group. | 2.4407 (2.1437)
  Day 15: number analyzed (Participants) | 6 | 6 | 6 | 5 | 0 | 0
  Day 15 | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.0000 (0.0000) | 5.4320 (2.6999) |  |
  Day 17: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 5
  Day 17 |  |  |  |  | 0.0000 (NA) — Standard deviation was not applicable as only one participant was evaluable for this reporting group. | 0.3980 (0.8900)
  Day 22: number analyzed (Participants) | 6 | 6 | 6 | 5 | 0 | 0
  Day 22 | 0.0000 (0.0000) | 0.0000 (0.0000) | 0.5478 (0.8613) | 7.1622 (2.7936) |  |

12. Secondary Outcome: Change From Baseline in Serum Concentration for Total LCAT Activity
Description: Lecithin-cholesterol acyltransferase (LCAT) is a plasma enzyme secreted by the liver. Serum LCAT activity was estimated to provide an alternative measure to LCAT mass in establishing the relationship between pharmacokinetics and pharmacodynamics of MEDI6012. Change in LCAT activity from baseline (pre-dose of each dose) to post doses was reported (concentration at Days 8, 15, and 22 for Cohorts 1 to 3 and placebo; Concentration at Days 3, 10, and 17 for Cohort 4 and placebo IV push arm).
Time Frame: as for outcome 11
Population: PK population included all participants in the as-treated population who had at least one detectable LCAT serum concentration measurement. LCAT activity at Day 3 and Day 17 were not collected for Cohort 4. The overall number of participants analyzed denotes the number of participants evaluated specific for this outcome measure.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Placebo | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Placebo IV Push | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 1 | 7
μg/mL
  Day 8: number analyzed (Participants) | 5 | 6 | 4 | 2 | 0 | 0
  Day 8 | 0.2046 (0.3035) | 0.0282 (0.9432) | 0.6710 (0.8715) | 0.9720 (0.7029) |  |
  Day 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 7
  Day 10 |  |  |  |  | 0.0000 (NA) — Standard deviation was not applicable as only one participant was evaluable for this reporting group. | 0.5503 (0.5960)
  Day 15: number analyzed (Participants) | 6 | 6 | 6 | 5 | 0 | 0
  Day 15 | -0.1467 (0.8494) | 0.1700 (0.7582) | 0.2418 (0.9939) | 1.1188 (0.7320) |  |
  Day 22: number analyzed (Participants) | 4 | 6 | 5 | 0 | 0 | 0
  Day 22 | 0.4983 (0.3355) | -0.1617 (0.7031) | 0.0824 (1.0816) |  |  |

13. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of MEDI6012
Description: The maximum observed serum concentration following the first and third dose of MEDI6012 was reported.
Time Frame: Day 1 end of infusion to Day 8 predose for Cohorts 1 to 3; Day 1 end of infusion to Day 3 predose for Cohort 4; Cmax following the third dose: Day 15 end of infusion to Day 71 for Cohort 1 to 3; Day 10 end of infusion to Day 65 for Cohort 4.
Population: PK population included all participants in the as-treated population who had at least one detectable LCAT serum concentration measurement. The overall number of participants analyzed denotes the number of participants evaluated specific for this outcome measure.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 5 | 5
μg/mL
  Dose 1 | 9.17 (3.27) | 27.5 (7.78) | 83.7 (27.7) | 75.1 (14.6)
  Dose 3 | 9.63 (3.5) | 27.1 (5.37) | 94.7 (33.1) | 28.5 (6.89)

14. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of MEDI6012
Description: The time to reach the maximum observed serum concentration following the first and third dose of MEDI6012 was reported.
Time Frame: Day 1 end of infusion to Day 8 predose for Cohorts 1 to 3; Day 1 end of infusion to Day 3 predose for Cohort 4; Tmax following the third dose: Day 15 end of infusion to Day 71 for Cohort 1 to 3; Day 10 end of infusion to Day 65 for Cohort 4.
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 6 | 5
Hours
  Dose 1 | 0.0417 (0.00) | 0.0417 (0.00) | 0.0417 (0.00) | 0.000696 (0.00)
  Dose 3 | 14.0417 (0.00) | 14.0417 (0.00) | 14.0417 (0.00) | 9.00070 (0.00)

15. Secondary Outcome: Accumulation Ratio (Rac) of MEDI6012
Description: The accumulation ratio (Rac) is defined as the ratio of accumulation of a study drug going from a single dose to steady state with repeated administration. Accumulation ratio was reported on the basis of maximum concentration (ARC max) and area under the concentration-time curve (ARAUC).
Time Frame: Day 1 end of infusion to Day 8 predose for Cohorts 1 to 3; Day 1 end of infusion to Day 3 predose for Cohort 4; The Rac following third dose: Day 15 end of infusion to Day 71 for Cohort 1 to 3; Day 10 end of infusion to Day 65 for Cohort 4.
Population: PK population. The Rac was not calculated for Cohort 4 as the first dose regimen (300 mg loading dose follow by 2nd dose given 48 hours later, therefore NCA was not performed for Dose 1) are different from 3rd dose (100 mg). The overall number of participants analyzed denotes the number of participants evaluated specific for this outcome measure.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 6 | 7
Ratio
  ARCmax: number analyzed (Participants) | 6 | 6 | 5 | 0
  ARCmax | 1.09 (0.214) | 1.01 (0.112) | 1.02 (0.177) |
  ARAUC: number analyzed (Participants) | 1 | 4 | 5 | 0
  ARAUC | 0.897 (NA) — Standard deviation was not applicable as only one participant was evaluable for this reporting group. | 1.16 (0.0982) | 1.21 (0.169) |

16. Secondary Outcome: Terminal Half-life (t1/2) of MEDI6012
Description: The t1/2 is the time measured for the serum concentration to decrease by one half after the third dose of MEDI6012.
Time Frame: The t1/2 following third dose: Day 15 end of infusion to Day 71 for Cohort 1 to 3; Day 10 end of infusion to Day 65 for Cohort 4.
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 1 | 5 | 5 | 4
Days | 2.7 (NA) — Standard deviation was not applicable as only one participant was evaluable for this reporting group. | 1.79 (0.374) | 2.52 (0.702) | 2.6 (0.942)

17. Secondary Outcome: Area Under the Concentration Time Curve to Last Measurable Time Point (AUClast) of MEDI6012
Description: The area under the concentration time-curve to the last measured concentration after the third dose of MEDI6012 was reported.
Time Frame: Day 1 end of infusion to Day 8 predose for Cohorts 1 to 3; Day 1 end of infusion to Day 3 predose for Cohort 4; AUClast following the third dose: Day 15 end of infusion to Day 71 for Cohort 1 to 3; Day 10 end of infusion to Day 65 for Cohort 4.
Population: PK population. The AUClast was not reported following first dose in Cohort 4 since NCA was not performed due to dosing period was only 48 hrs. The overall number of participants analyzed denotes the number of participants evaluated specific for this outcome measure.
Measure: Mean (Standard Deviation); unit: µg*day/mL
Arm/Group | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 6 | 5
µg*day/mL
  Dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0
  Dose 1 | 10.9 (10.1) | 35.2 (17.8) | 152 (50.5) |
  Dose 3: number analyzed (Participants) | 6 | 6 | 5 | 5
  Dose 3 | 8.98 (5.61) | 48.3 (23.6) | 205 (63.7) | 38.6 (21.9)

18. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies for MEDI6012
Description: Participants with positive serum antibodies to MEDI6012 were reported.
Time Frame: For Cohorts 1 to 3 and Placebo arm: Pre-dose on Days 1 and 15, and on Days 29, 43, and 71; For Cohort 4 and Placebo IV push arm: Pre-dose on Days 1 and 10, and on Days 24, 38, and 66.
Population: Immunogenicity population included all participants in the as-treated population who had at least one serum sample for immunogenicity testing
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cohort 1: MEDI6012 40 mg | Cohort 2: MEDI6012 120 mg | Cohort 3: MEDI6012 300 mg | Placebo IV Push | Cohort 4: MEDI6012 IV Push
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 1 | 7
Participants
  ADA positive at baseline | 0 | 0 | 0 | 0 | 0 | 0
  ADA positive post-baseline | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline (Day 1) to Day 56 after last dose of study drug (Day 66 for Cohort 4 and Placebo IV push arm and Day 71 for Cohorts 1 to 3 and placebo arm).
Groups:
- Placebo: Description (Arm-group)
Arm/Group | Placebo | MEDI6012 40 mg | MEDI6012 120 mg | MEDI6012 300 mg | Placebo IV Push | MEDI6012 IV Push
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/1 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 0/6 | 0/1 | 0/7
Other Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 3/6 | 4/6 | 0/1 | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | MEDI6012 40 mg (N=6) | MEDI6012 120 mg (N=6) | MEDI6012 300 mg (N=6) | Placebo IV Push (N=1) | MEDI6012 IV Push (N=7)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | MEDI6012 40 mg (N=6) | MEDI6012 120 mg (N=6) | MEDI6012 300 mg (N=6) | Placebo IV Push (N=1) | MEDI6012 IV Push (N=7)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2017-07-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT03004638/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT03004638/SAP_001.pdf